CLINICAL TRIAL: NCT06399887
Title: Evaluation of the Effectiveness of Dynamic Neuromuscular Stabilization Training in Children With Lower Urinary Tract Dysfunction: a Pilot Study
Brief Title: Investigation of the Effectiveness of Different Interventions for Lower Urinary Tract Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Emine Nacar, Research Assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-06/12
Record Dates: First submitted 2024-04-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Lower Urinary Tract Symptoms; Biofeedback; Pelvic Floor
Keywords: Children; lower urinary tract dysfunction; dynamic neuromuscular stabilization; biofeedback; pelvic floor rehabilitation
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Exercise; Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I : Dynamic neuromuscular stabilization exercise training (Active Comparator): Group I
  • dynamic neuromuscular stabilization exercise training
  * 45 minute/ 3 sessions/ week
  * 12 weeks
  Interventions: Other: Exercise
- Group II : Biofeedback training (Active Comparator): Group II
  • biofeedback training
  * 20 minute/ 1 sessions/ week
  * 12 weeks
  Interventions: Other: Biofeedback
- Group III : Dynamic neuromuscular stabilization exercise training + biofeedback training (Active Comparator): Group III
  * dynamic neuromuscular stabilization exercise training
    * 45 minute/ 3 sessions/ week
    * 12 weeks
  * biofeedback training
    * 20 minute/1 sessions/week
    * 12 weeks
  Interventions: Other: Exercise; Other: Biofeedback

INTERVENTIONS:
Other: Exercise — All patients in these groups are taught diaphragmatic breathing, which is the basis for DNS, and are asked to maintain it throughout the exercises. The DNS protocol includes a 5-minute warm-up, 40 minutes of DNS exercises (10 minutes for each of the 4 different body parts) and breathing exercises. The DNS exercises included diaphragmatic breathing, Baby Rock, Roll Over, Lying on the Side, Sitting Down, Sitting Upright, Tripod, Kneeling, Squatting, Prone, and Pull Up (CGU). The focus of the first week is to teach and practice basic DNS exercises.
  Arms: Group I : Dynamic neuromuscular stabilization exercise training; Group III : Dynamic neuromuscular stabilization exercise training + biofeedback training
Other: Biofeedback — Patients in Group II and Group III will be trained in animated CP using the Aymed Medical Locum Wireless System v.2.69.0.12 device. During CP, 10-second contraction and 30-second relaxation cycles are maintained throughout the animated game. Each session will last approximately 20 minutes. The training protocol will consist of a total of 12 sessions of 20 minutes per week for 3 months.
  Arms: Group II : Biofeedback training; Group III : Dynamic neuromuscular stabilization exercise training + biofeedback training

SUMMARY:
Lower urinary tract dysfunction (LUTD) is present in 2-40% of healthy children. If left untreated, it can lead to health problems such as recurrent urinary tract infections, vesicoureteral reflux and chronic renal failure. Pelvic floor physiotherapy is a globally accepted treatment for adults and children. In addition to locomotor skills, functional exercises such as motor control, core stability and balance training are important to support toilet training. Dynamic Neuromuscular Stabilization (DNS), a current stabilization approach, is a neurophysiological rehabilitation strategy based on developmental kinesiology, using ontogenetic models to both diagnose and treat dysfunction in the locomotor system in infants and adult patients. Today, DNS is successfully used in the rehabilitation of various neurological, musculoskeletal, pediatric and sports injuries. However, there are no studies in the literature examining the effectiveness of DNS training in children diagnosed with LUTD. The aim of this study was to evaluate the effectiveness of DNS training in children diagnosed with LUTD and to compare it with EMG-Biofeedback treatment method. The children participating in the study will be randomly divided into 3 groups. Children in Group I will exercise 3 days a week for 45 minutes according to DNS principles. Children in Group II will receive EMG Biofeedback training 1 day a week. Children in Group III will receive EMG-Biofeedback training 1 day a week in addition to exercises with DNS principles 3 days a week. In the study, data on symptoms, demographic data of the individuals before treatment and at 4th week, 8th week and 12th week after treatment will be obtained from each child participating in the study through a questionnaire, symptoms related to voiding disorder and urinary incontinence with Dysfunctional Voiding and Incontinence Scoring System (DVISS), activation of deep trunk muscles with Stabilizer Pressure Biofeedback Unit, urine flow curve and voiding parameters of the patients with uroflowmeter application will be evaluated. Kruskal-Wallis analysis of variance will be used to compare the three groups in terms of variables. Wilcoxon signed-rank test will be used to analyze the statistical significance of the difference between all values before and after treatment. For all results, p<0.05 will be considered as significance level.

DETAILED DESCRIPTION:
The sample of the study will consist of children between the ages of 6-15 years who were admitted to Malatya Inönü University Turgut Özal Medical Center Pediatric Urodynamics/Urotherapy Unit and diagnosed with LUTD by a pediatric nephrology specialist. Inclusion criteria: Being between the ages of 6-15 years, having a normal neurologic examination, being diagnosed with LUTD, having a DVISS of 8.5 and above, not having received any medication or other treatment for enuresis before. Exclusion criteria were as follows: patients with primary nocturnal enuresis, patients with uncontrolled systemic disease, patients with neurologic disease (muscle disease, epilepsy, etc.), patients with inflammation of the vagina, anus and urinary tract, patients with febrile illness or active urinary tract infection, presence of underlying psychological causes, presence of mental retardation, inability to comply with treatment. Children who meet the inclusion criteria will be included in the study by non-probability random sampling method. The inclusion of the three clusters formed according to the registration number of the Pediatric Urodynamics/Urotherapy Unit will be determined by lottery method. After the children and their parents/guardians who meet the inclusion criteria are informed about the study content, they will be asked to sign the informed consent forms for the child and the informed consent forms for the parents/guardians if they agree to participate in the study.

The individuals participating in the study will be divided into 3 groups. Children in Group I will exercise according to DNS principles 3 days a week for 12 weeks, with sessions of 45 minutes. Children in Group II will receive animated EMG biofeedback training with the Aymed Medikal Locum Wireless System v.2.69.0.12 device. For animated biofeedback application, two electrodes will be placed at 3 and 9 o'clock in the perineum region and 1 reference electrode will be placed on the inner side of the thigh (42). The training protocol will be applied once a week for a total of 12 sessions for 3 months. In addition to exercises with the DNS principle 3 days a week, the children in Group III will receive biofeedback training with animation once a week with the Aymed Medikal Locum Wireless System v.2.69.0.12 device for a total of 3 months. Demographic data of the individuals participating in the study will be obtained through a questionnaire from each child participating in the study. The questions in the questionnaire are personal information of the child, toilet training age, frequency of urinary tract infections, whether they have received treatment for urinary incontinence before, whether they have chronic constipation, whether their parents have a history of urinary incontinence at a young age and some personal information specific to the parents.

The Dysfunctional Voiding and Incontinence Scoring System (DVISS) will be used for symptoms of voiding dysfunction and urinary incontinence. The DVISS is a 13-item questionnaire. It originally includes 14 questions about symptoms and 1 question about quality of life. In the scoring system developed by Akbal et al. for the pediatric population and adapted to Turkish, there are 13 symptom and 1 quality of life question.

Evaluation of uroflowmeter parameters will be performed with the uroflowmeter application of the Aymed Medikal Locum Wireless System v.2.69.0.12 EMG device and the urine flow curve and voiding parameters of the patients will be evaluated. These parameters are maximum flow rate, time to reach maximum flow, mean flow rate, voiding volume and voiding time. In our study, urine volume of 100 ml or more will be considered valid. Evaluation of deep trunk muscles (transversus abdominis, multifidus and deep neck flexors) will be performed with the Stabilizer Pressure Biofeedback Unit (Chattanooga Stabilizer, USA). Before the test, each participant will be taught how to contract the transversus abdominis muscle with the corset method in the supine and quadripedal position and how to contract the multifidus muscle in the supine position. Measurements will be made for 10 seconds and 3 repetitions, three measurements will be recorded and averaged. For the measurement of the deep neck flexors, the patients will first be taught the correct craniocervical flexion movement without activation of the superficial muscles. The change in pressure will be recorded and the highest value from 3 trials will be taken. Individuals will be evaluated before treatment, at 4 weeks, 8 weeks and 12 weeks after treatment. The aim here is to measure how long it takes to show the effectiveness of the treatment(s) applied and to determine whether the treatments are superior in terms of time.

ELIGIBILITY:
Inclusion Criteria:

* - Normal growth and development,
* Absence of a known psychological or behavioural disorder and interactive communication problems or chronic drug use related to these diseases.
* Normal mental, motor development, and neurological examination findings without any neuro-motor system abnormalities,
* Absence of any current and/or past congenital anomalies and abnormal ultrasonography (USG) examination findings in the kidney and urinary tract,
* Dysfunctional Voiding and Incontinence Symptoms Score Questionnaire (DVISS) score above 8.5 points

Exclusion Criteria:

* - Skin findings that may be related to occult spinal dysraphism in the lumbosacral region examination,
* In the uroflowmetry (UFM) test;
* Voided volume (VV) is less than 100 mL and/or below 50% or above 115% of expected bladder capacity (EBC)

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Lower urinary tract symptom score | 12 weeks
  The DVISS recommended by the ICCS will be used for the evaluation of lower urinary tract function. This questionnaire, which has Turkish validity and reliability, consists of 13 symptoms and 1 quality of life question. The total score varies between 0 and 35. An increase in the total score indicates an increase in symptoms. It has a cut-off value of 8.5 and 90% specificity and sensitivity in detecting the presence of bladder bowel dysfunction and LUTD.
Post-voiding residual urine | 12 weeks
  PVR and rectal diameter assessment of the children will be performed by the same person in the same unit with a Logiq P9 USG Device (GE Healthcare, USA) within the first 5 minutes after the UFM test. Pelvic USG is performed with a 5 mHz low frequency convex USG probe. The convex probe is placed 1-2 cm above the symphysis pubis and images of the bladder are taken in the transverse and sagittal axes. PVR will be calculated using the ellipsoid formula based on measurements of the bladder at its maximal diameters as follows: anteroposterior diameter x transverse diameter x longitudinal diameter x 0.52. For children aged 4-6 years, a single PVR >30 ml or >21% of BC, repeat PVR >20 ml or >10% of BC; for children aged 7-12 years, a single PVR >20 ml or >15% of BC, repeat PVR >10 ml or >6% of BC is considered significantly high.
Flow curve type | 12 weeks
  The urine flow curve will be interpreted by a pediatric nephrologist according to the pattern of the curve obtained from the voiding test. According to ICCS recommendations, five different types of voiding curves can be seen on the uroflowmeter. These are bell, tower, plateau, staccato and fractional and only the bell-shaped voiding curve is considered normal. The presence or absence of these parameters and voiding curves within normal limits provides important objective information about voiding dysfunctions.
Deep trunk muscle strength | 12 weeks
  Assessment of the deep trunk muscles, especially the Transversus Abdominis (TrA) and deep neck flexors (DNF) will be performed using the Stabilizer Pressure Biofeedback Unit (Chattanooga Stabilizer).
Voiding volume | 12 weeks
  Voiding volume, one of the uroflowmeter parameters, will be performed using the Intelligent System UFM Device (Serial No: 18020004-02) (Uroscan Plus Inoflow Intelligent UFM Device, Aymed, Medical Technology, Turkey).
Voiding time | 12 weeks
  Voiding time, one of the uroflowmeter parameters, will be performed using the Intelligent System UFM Device (Serial No: 18020004-02) (Uroscan Plus Inoflow Intelligent UFM Device, Aymed, Medical Technology, Turkey).
Maximum flow rate | 12 weeks
  Maximum flow rate, one of the uroflowmeter parameters, will be performed using the Intelligent System UFM Device (Serial No: 18020004-02) (Uroscan Plus Inoflow Intelligent UFM Device, Aymed, Medical Technology, Turkey).
Time to reach maximum flow | 12 weeks
  Time to reach maximum flow, one of the uroflowmeter parameters, will be performed using the Intelligent System UFM Device (Serial No: 18020004-02) (Uroscan Plus Inoflow Intelligent UFM Device, Aymed, Medical Technology, Turkey).
Average flow rate | 12 weeks
  Average flow rate, one of the uroflowmeter parameters, will be performed using the Intelligent System UFM Device (Serial No: 18020004-02) (Uroscan Plus Inoflow Intelligent UFM Device, Aymed, Medical Technology, Turkey).

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Suner Keklik, Assoc. Prof., Study Director — Cumhuriyet University; Ahmet Taner Elmas, Prof., Study Director — İnönü University
Locations (1):
- Department of Pediatric Nephrology, Inonu University Faculty of Medicine, Turgut Özal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No